CLINICAL TRIAL: NCT02865408
Title: Enhancing the Anabolic Effect of Nutrition in Critically Ill Patients by Administering Exogenous Amino Acids
Brief Title: Amino Acid Nutrition in the Critically-ill
Acronym: AA-ICU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arnold Kristof (Other)
Responsible Party: Sponsor-Investigator, Arnold Kristof, Doctor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4738
Record Dates: First submitted 2015-07-07; First posted 2016-08-12 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; Inflammation; Malnutrition
Keywords: Amino acids; critically-ill; catabolic; nutrition; anabolic
MeSH Terms: conditions — Critical Illness; Inflammation; Malnutrition | interventions — Peptamen; Enteral Nutrition; Amino Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Peptamen 1.5% via enteral only (Active Comparator): Study patients in this group will be prescribed 1.0 g/kg/d of protein using standard EN Peptamen 1.5%. Based on current compliance or tolerance statistics, investigators expect patients to only receive 50-60% of these prescribed doses; effective protein intake will therefore be approximately 0.5-0.6 g/kg/d
  Interventions: Dietary Supplement: Peptamen 1.5% via enteral
- Group 2: Prosol 20% IV to 1.75g/kg/day (Active Comparator): Patients in group 2 will receive the same enteral feeding as group 1 (Peptamen 1.5) but in addition will receive sufficient intravenous amino acid supplements (Prosol 20%) to achieve an effective fixed dose of 1.75 g/kg/d
  Interventions: Dietary Supplement: Peptamen 1.5% via enteral; Dietary Supplement: Prosol 20% IV to 1.75g/kg/day
- Group 3: Prosol 20% IV to 2.5g/kg/day (Active Comparator): Patients in this group will receive intravenous amino acids (Prosol 20%) in addition to standard enteral Peptamen 1.5% to achieve an effective protein intake of 2.5 g/kg/day.
  Interventions: Dietary Supplement: Peptamen 1.5% via enteral; Dietary Supplement: Prosol 20% IV to 2.5g/kg/day

INTERVENTIONS:
Dietary Supplement: Peptamen 1.5% via enteral — Study patients in this group will be prescribed 1.0 g/kg/d of protein using standard enteral Peptamen 1.5%. Based on current compliance or tolerance statistics, investigators expect patients to only receive 50-60% of these prescribed doses; effective protein intake will therefore be approximately 0.5-0.6 g/kg/d.
  Other Names: Enteral feeding with Peptamen 1.5%
Dietary Supplement: Prosol 20% IV to 1.75g/kg/day — Patients in group 2 will receive Peptamen 1.5% but in addition, will receive sufficient intravenous amino acid supplements (Prosol 20%) to achieve an effective fixed dose of 1.75 g/kg/day.
  Other Names: Enteral feeding with Peptamen 1.5% plus Prosol 20%
  Arms: Group 2: Prosol 20% IV to 1.75g/kg/day
Dietary Supplement: Prosol 20% IV to 2.5g/kg/day — Patients in this group will receive intravenous amino acids, Prosol 20% in addition to standard enteral Peptamen 1.5% to achieve an effective protein intake of 2.5 g/kg/d.
  Other Names: Enteral feeding with Peptamen 1.5% plus Prosol 20%
  Arms: Group 3: Prosol 20% IV to 2.5g/kg/day

SUMMARY:
Enhancing the anabolic effect of nutrition in critically ill patients by administering exogenous amino acids.

DETAILED DESCRIPTION:
Critically-ill patients admitted to the intensive care unit are invariably catabolic and are commonly undernourished. Previous observational studies indicate that increased dietary administration of protein or essential amino acids might be associated with improved clinical outcomes. The investigators propose that the parenteral supplementation of intravenous amino acids in critically-ill patients will restore anabolic processes and that anabolism is associated with molecular markers of amino acid sensing and protein synthesis. The results from this study will establish biomarkers of anabolism (i.e., nutritional success) that can be used in future clinical trials on the use of amino acid supplementation in the critically-ill.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated adult patients (>18 years old) admitted to ICU with an expected ICU dependency (alive and need for mechanical ventilation
* Vasopressor therapy, or mechanical circulatory support) at the point of screening of an additional 3 days, as estimated by the treating physician.

Exclusion Criteria:

* Patients who are moribund (expected death within 48 hours)
* Expected to have life-sustaining treatments withdrawn in the next 3 days
* Those with a contraindication to enteral nutrition (EN)
* Already on parenteral nutrition (PN)
* Those with acute fulminant hepatitis or severe chronic liver disease (Child's class C)
* Patients on extracorporeal membrane oxygenation or carbon dioxide removal* Patients with organ transplantation
* Those with a broncho-pleural fistula
* Patients with documented allergies to any of the study nutrients or its excipients will be excluded.
* Patients requiring continuous renal replacement therapy or extracorporeal membrane oxygenation are excluded due to inability to accurately measure protein turnover.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Whole body protein balance | 0 and 48 hours
  Primed continuous infusions of stable isotope tracers will be applied to assess dynamic changes in whole body and hepatic protein metabolism (i.e., protein breakdown, amino acid oxidation, protein synthesis, total protein, albumin and fibrinogen synthesis) before 48 hours after beginning the intervention. During the period of isotope infusion, nutrition will be held constant. A positive protein balance (difference between protein synthesis and protein breakdown) will be used as an indicator of whole body anabolism. All isotopes will be purchased from CDN Laboratories (Montreal, Canada). Sterile solutions will be tested to be free of pyrogens. Before beginning each experiment blood and expired air samples will be collected to determine baseline enrichments of [1-13C]-ketoisocaproate ([1-13C]-KIC), [6,6-2H2]glucose, L-[2H5]phenylalanine and expired 13CO2. Retention of H13CO3- in the bicarbonate pool will be measured in each patient using the approach of Kien.

SECONDARY OUTCOMES:
Synthesis rates of hepatic secretory proteins (the total plasma protein pool, albumin, fibrinogen in %/d) | 0 and 48 hours
  This will be measured from the rates of incorporation of L-[2H5] phenylalanine into the proteins using plasma very low density lipoprotein apolipoprotein-B100 (VLDL-apoB-100) isotopic enrichment at plateau to represent the isotopic enrichment of the phenylalanine precursor pool from which the liver synthesizes the other plasma protein. A priming dose of L-[2H5]phenylalanine (4 μmol/kg, iv) will be given followed by a six-hour infusion at 0.10 μmol/kg/min. At baseline, 3 hours, 4 hours, 5 hours, and 6 hours thereafter blood will be drawn, immediately transferred into pre-chilled tubes containing Na2EDTA and a protease inhibitor cocktail of sodium azide, merthiolate and soybean trypsin inhibitor, then centrifuged and stored at -70ºC for later analysis. 10 ml blood will be required for secretory protein synthesis studies.
Biomarker of amino acid restriction or repletion - ELISA (pg/ml) | 0, 12, 24, 36, 48, 72 hours
  Blood (one 4-ml tube per sample) will be collected at baseline, then every 12 hours in the first 48 hours, and 72 hours post initiation of amino acid administration. Measures of amino acid-sensitive inflammation include the following: serum C-reactive protein and interleukin-6.
Biomarker of amino acid restriction or repletion - mRNA detection (copy number/ml) | 0, 12, 24, 36, 48, 72 hours
  Blood (one 2.5-ml tube per sample) will be collected at baseline, then every 12 hours in the first 48 hours, and 72 hours post initiation of amino acid administration. Using Pax-gene tubes, peripheral blood mononuclear cell (PBMC) mRNA will be isolated for detection of interleukin-6 and c-reactive protein gene expression.
Biomarker of amino acid restriction or repletion - protein levels (fold increase in Western blot band density) | 0, 12, 24, 36, 48, 72 hours
  Blood (one 4 ml cell separator tube per sample) will be collected at baseline, then every 12 hours in the first 48 hours, and 72 hours post initiation of amino acid administration. Measures of amino acid-sensitive cell signaling in peripheral blood mononuclear cells include: phospho- p70 S6 kinase, phospho-S6, or phospho-eiF2α by Western blot.
Metabolic Substrates (micromolar) | 0, 24, 36, 48, 72 hours
  Plasma amino acids and markers of oxidative stress (glutathione, cysteine, related sulfhydryl) by liquid chromatography tandem mass spectroscopy. Blood will be collected at baseline, then at 24, 48, and 72 hours initiation of amino acid administration.
Resting Energy Expenditure (kcal) | 0 and 48 hours
  Investigators will measure resting energy expenditure by indirect calorimetry at the 5 hour time point of each tracer protocol (Baseline and 48 h after initiation of amino acid administration. This will permit comparison of actual energy expenditure with that estimated by weight-based nomogram used for nutritional dosing.

OTHER OUTCOMES:
ICU length of stay | 72 hours to 1 year
  Duration of ICU admission in days.
Hospital length of stay | 72 hours to 1 year
  Duration of ICU admission in days.
Ventilator-free days in ICU | 72 hours to 1 year
  Duration of stay in ICU off mechanical ventilation.
Hospital-acquired infections. | 72 hours to 1 year
  Number of hospital-acquired infections during the hospital admission.
Mortality | 72 hours to 1 year
  Death in hospital (binary value for dead or alive).

CONTACTS AND LOCATIONS:
Overall Officials: Arnold S Kristof, MDCM, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kristof AS, Hong M, Boufaied N, Tousson-Abouelazm N, Dandamudi S, Joung KB, Hatzakorzian R, Port M, Campisi G, Piccirillo CA, Fonseca GJ, Ding J, Heyland DK, Labbe DP, Wykes L, Schricker T. Biological responses during high-dose protein nutrition in the critically ill: a randomized controlled trial. Am J Clin Nutr. 2025 Aug;122(2):612-623. doi: 10.1016/j.ajcnut.2025.05.025. Epub 2025 Jun 26. PMID 40617772
- [Derived] Omiya K, Sato H, Sato T, Wykes L, Hong M, Hatzakorzian R, Kristof AS, Schricker T. Albumin and fibrinogen kinetics in sepsis: a prospective observational study. Crit Care. 2021 Dec 17;25(1):436. doi: 10.1186/s13054-021-03860-7. PMID 34920728